CLINICAL TRIAL: NCT03628274
Title: Diagnosis and Definition of Local Involvement of Musculoskeletal Tumors: Assessment of Ultra-high Field MRI Exploration Contribution
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-39; 2018-A00925-50 (Registry Identifier: ID RCB)
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Magnetic Resonance Imaging (RMI) 7 Tesla (Experimental)
  Interventions: Device: Magnetic Resonance Imaging (MRI) 7 Tesla; Device: Magnetic Resonance Imaging (MRI) 1,5 Tesla

INTERVENTIONS:
Device: Magnetic Resonance Imaging (MRI) 7 Tesla — An MRI performed as part of the project
Device: Magnetic Resonance Imaging (MRI) 1,5 Tesla — An MRI performed as part of the care

SUMMARY:
Sarcomas are aggressive malignant tumors issued from mesenchymatous cells. Their curative treatment is mainly surgical, especially in soft tissue sarcomas, which are mostly localized in limbs. Surgical margins remain a major prognosis factor and are directly linked to recurrence risk. Curative surgery applies resection margins removing healthy tissue surrounding the tumor and is meticulously planned thanks to tight cooperation between expert surgeons and radiologist, based on pre-operative Magnetic resonance imaging(MRI). Resection planning optimizes chances to perform a safe carcinological resection procedure sparing these structures. Resection planning is based upon conservation (or sacrifice) of anatomic compartments limited by fascia and routine MRI might also be outdated in some cases to predict whether the fascia is involved in the tumor or not. Such uncertainties complexify the surgical procedure, lead to unnecessary healthy tissue sacrifices and increase functional impairments, which can be significant. A new MRI offering higher spatial resolution could allow tumoral satellites, previously undetected on conventional MRI, which might explain some of the observed recurrences. Ultra-high field MRI, considered as harmless and without pharmaceutical agent injection, could bring benefits to tumoral extension comprehension and should be considered as a breakthrough in medical oncology field. This is particularly true in soft tissue sarcoma pathology field, where the only curative treatment to date remains surgery.

It will be propose in this project to determine the contribution of ultra-high field MRI in Soft tissue sarcomas management and to evaluate for the first time the potential superiority of 7 Tesla imaging over routine MRI through usual data comparison in 20 patients between 1,5Tesla and 7 Tesla MRI.

ELIGIBILITY:
Inclusion Criteria:

* Major patients
* All patients with soft-tissue sarcoma
* Patients agreeing to participate in the study and having signed a consent

Exclusion Criteria:

* Patients with a contraindication to MRI will be excluded: Claustrophobia, metallic foreign bodies, cardiac pacemakers, implantable chamber. There is no known additional risk for 7Tesla MRI scanning. The same contraindications as those of conventional MRI prevail.
* Patients with bone-component sarcomas will be excluded in order to have a homogeneous group of tumors localized only in the soft tissues (and simpler analysis in high-field MRI because of the risk of artifacts related to bone).
* Intermediate malignancies will be excluded for the same reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
A subjective score of suspicion of the image defined by the Lickert scale | 24 months
  the invaded anatomical structures are evaluated by observation of images matched at the Lickert scale. It's based on a five stage Likert scale (0: formally benign, 1: probably benign, 2: undetermined, 3: probably malignant, 4: formally malignant).

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Director, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No